CLINICAL TRIAL: NCT02856334
Title: Psychosocial Factors and Central Sensitization in Chronic Pelvic Pain
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Rafael Torres Cueco, PT, University of Valencia
Other Study IDs: 0117
Record Dates: First submitted 2016-07-20; First posted 2016-08-04 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-08

CONDITIONS: Pelvic Pain; Vulvodynia; Pudendal Neuropathy
Keywords: chronic pelvic pain; vulvodynia; pelvic pain; psychosocial factors; central sensitization
MeSH Terms: conditions — Pelvic Pain; Vulvodynia; Pudendal Neuralgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- Chronic pelvic pain: Women with chronic pelvic pain
- Control group: Healthy women

SUMMARY:
The purpose of this study is to determine if the psychosocial factors in women with chronic pelvic pain are predisposing, precipitant or maintenance factors, and relate these factors with central sensitization and dysfunctional pain.

DETAILED DESCRIPTION:
This study pretends clarify the psychosocial factors presents in women with chronic pelvic pain, and determine if this factors are predisposing, precipitant or of maintenance, through an interview and a series of validated questionnaires. In addition, these findings will be related to the presence of central sensitization, as measured by quantitative sensory testing.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 55 years
* Chronic pelvic pain diagnosis, defined as persistent pain in pelvis related structures
* Pain duration ≥6 months
* Average pain intensity ≥3/10 in NRS during the previous week
* To understand the objectives of the study

Exclusion Criteria:

* Suspicion or knowledge of current organic pathology that requires medical or surgical treatment
* Pain as a consequence of surgery known
* Pending litigation or financial compensation
* Psychiatric disorders: major depression, bipolar syndrome, etc ..
* Cognitive difficulties
* Not sign the informed consent

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women with chronic pelvic pain
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Interview on psychosocial factors | Day 1

SECONDARY OUTCOMES:
Survey of Pain Attitudes-35 (SOPA-35) | Day 1
Multidimensional Pain Inventory (MPI) - Interference Scale | Day 1
Oswestry Disability Index | Day 1
Hospital Anxiety and Depression Scale (HADS) | Day 1
Pain Catastrophizing Scale | Day 1
Coping Strategies Questionnaire (CSQ) | Day 1
Tampa Scale for Kinesiophobia (TSK) -11 | Day 1
Neurophysiology of pain questionnaire (NPQ) | Day 1
Female Sexual Function Index (FSFI) | Day 1
Patient Specific Functional Scale (PSFS) | Day 1
Patient Health Questionnaire (PHQ) | Day 1
Quantitative Sensory Testing-Pain Pressure Threshold (PPT) | Day 2
  in kg/s
Quantitative Sensory Testing-Temporal Summation (TS) | Day 2
  in kg/s
Quantitative Sensory Testing-Conditioned Pain Modulation (CPM) | Day 2
  in kg/s

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Torres-Cueco, Principal Investigator
Locations (2):
- Spain (2):
  - Rafael Torres, Valencia, Valencia
  - Valencia, Valencia